CLINICAL TRIAL: NCT03023267
Title: Open Randomized Study on the Effect of Applying Music Therapy by Therapist in the Neonatal Intensive Care Unit (NICU).
Brief Title: The Contribution of Parent-infant Interaction While Singing During Kangaroo Care, on Preterm-infants' Autonomic Stability and Parental Anxiety Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Shmuel Arnon, Senior Neonatologist, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0283-15-MMC
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: PreTerm Birth; Stress Reaction
MeSH Terms: conditions — Premature Birth; Fractures, Stress | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Applying music therapy with kangaroo care to mothers and fathers during their NICU hospitalization
  Interventions: Behavioral: Music therapy and Kangaroo care
- Control (Active Comparator): Applying only Kangaroo care to mothers and fathers during their stay in the NICU
  Interventions: Behavioral: Kangaroo Care alone

INTERVENTIONS:
Behavioral: Music therapy and Kangaroo care — Mother holding baby in skin to skin position while singing
  Arms: Interventional
Behavioral: Kangaroo Care alone — Mother holding baby in skin to skin position without singing
  Arms: Control

SUMMARY:
The current study will investigate the combination of the two modalities in a mixed-methods design, in order to provide comprehensive knowledge regarding the effects of family-centered MT during KC, on premature-infants' autonomic nervous system stability (measured by parasympathetic tone, physiological vital signs and behavioral states); Parents' anxiety levels; And parents' unique experiences of the intervention. Additionally, the study will analyze separately mothers and fathers to elucidate similar and different effects

DETAILED DESCRIPTION:
Premature infants and their parents are prone to high anxiety levels and a risk of experiencing trauma due to the preterm birth and its implications. Facing various emotional physical and neural high-risk factors may lead to continuous stress reactions in both the infant and parents, affecting their well being, the parent-infant relationship and the infant's medical state outcome. Attending to both infants' emotional and physiological needs of stability and comfort, as well as parents' support, can lead to an improvement in the premature infants' medical state and the parent-infant bonding process. Furthermore, reducing stress reaction facilitates perceptual memory and learning in premature infants. Two well established interventions in the neonatal care aiming to address the varied premature-family needs are Kangaroo care (KC) and Music Therapy (MT). Various research and clinical reports over the last three decades, regarding each modality, has shown beneficial effects in improvement and stabilization of infants' medical state, inclusion of parents in their infants' treatment and in facilitation of meaningful parent-infant interactions to promoting bonding patterns. However, a major lack of rigorous Randomized control studies presenting the clinical applications of MT techniques and methods in the NICU care exists, as well as only few research have positioned the parents in center of investigation, and/or presented their outcome and perspective. Accordingly, only few research have investigated the combination of MT and KC through an RCT. The current study will investigate the combination of the two modalities in a mixed-methods design, in order to provide comprehensive knowledge regarding the effects of family-centered MT during KC, on premature-infants' autonomic nervous system stability (measured by parasympathetic tone, physiological vital signs and behavioral states); Parents' anxiety levels; And parents' unique experiences of the intervention. Additionally, the study will analyze separately mothers and fathers to elucidate similar and different effects

ELIGIBILITY:
Inclusion criteria:

1. Preterm infants ≤ 37 weeks' gestation
2. Clinically stable preterm
3. Hearing confirmed by distortion product oto- acoustic emissions

Exclusion criteria:

1. Preterm infants treated with Central Nervous System (CNS) related medication (Luminal, Oxygen)
2. Infants with Intraventricular hemorrhage stage ≥ 3, Peri ventricular Leukomalacia
3. Parents refusal to participate

Ages: 4 Weeks to 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
parasympathetic tone | During intervention of music and\or kangaroo care which will carry on once during 32-36 weeks gestation and once at 3 months corrected age
  The electrocardiogram analogue signal from a cardiorespiratory monitor fed into a computer containing the Heart Rate Variability (HRV) software (ANSR1000 system Ansar, Inc., Philadelphia, Pennsylvania , USA). The analogue electrocardiogram signal is converted to digital values reflecting cyclic changes in the RR interval. The data is transformed into a waveform across a spectrum of various frequencies. Frequencies measured in hertz (1 Hz = 1 cycle/sec). Applied to variability, The high frequency (HF) power spectrum is in the frequency range of >0.15-1.80 Hz, which is predominately influenced by parasympathetic inputs.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grause, RD, Study Chair — Meir Medical Center
Locations (1):
- Neonatal Intensive Care Unit, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yakobson D, Arnon S, Gold C, Elefant C, Litmanovitz I, Beck BD. Music Therapy for Preterm Infants and Their Parents: A Cluster-Randomized Controlled Trial Protocol. J Music Ther. 2020 May 2;57(2):219-242. doi: 10.1093/jmt/thaa002. PMID 32112555